CLINICAL TRIAL: NCT00536198
Title: Symptom Onset Antidepressant Treatment for PMDD
Brief Title: Evaluating the Effectiveness of Sertraline in Treating Women With Premenstrual Dysphoric Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kimberly Yonkers, Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0609001839; R01MH072955 (NIH); DSIR 83-ATSO (Other Grant/Funding Number: National Institute of Mental Health)
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Premenstrual Dysphoric Disorder
Keywords: Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Dysphoric Disorder; Premenstrual Syndrome | interventions — Sertraline; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sertraline (Experimental): Participants will take sertraline that is dosed between 50 and 100 mgs during the symptomatic period. Women who report moderate to severe side effects will be allowed to reduce their dose to 25 mg of sertraline and to increase the dose at the next cycle unless rate-limiting side effects continue.
  Interventions: Drug: Sertraline
- Placebo (Placebo Comparator): Participants will take similar looking placebo during the symptomatic period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sertraline — 50 mg of sertraline will be taken at the onset of premenstrual symptoms through the first few days of menses. If a participant shows an insufficient response to this dose, the dose may be increased to 100 mg. Women who report moderate to severe side effects will be allowed to reduce their dose to 25 mg of sertraline and to increase the dose at the next cycle unless rate-limiting side effects continue.
  Other Names: Zoloft
  Arms: Sertraline
Drug: Placebo — 50 mg of placebo will be taken at the onset of premenstrual symptoms through the first few days of menses. If a participant shows an insufficient response to this dose, the dose may be increased to 100 mg.
  Other Names: Placebo, sugar pill
  Arms: Placebo

SUMMARY:
This study will evaluate the effectiveness of sertraline in reducing symptoms in women diagnosed with premenstrual dysphoric disorder.

DETAILED DESCRIPTION:
Premenstrual dysphoric disorder (PMDD) is a severe form of premenstrual syndrome (PMS). PMDD affects nearly 5 percent of menstruating women in the United States. This disorder is very disruptive and can affect a woman's performance at work and her relationships with friends and family. Symptoms typically occur 10 to 14 days before the start of a woman's period and dissipate soon after. Sadness, rapid changes in mood, anxiety, and irritability are common symptoms associated with PMDD. Sertraline is a selective serotonin reuptake inhibitor (SSRI) that has been approved by the U.S. Food and Drug Administration (FDA) to treat PMDD. This study will evaluate the effectiveness of sertraline in reducing symptoms in women diagnosed with PMDD.

All participants will begin this study by recording their symptoms for two complete menstrual cycles. At a baseline study visit, participants will then be randomly assigned to receive either sertraline or placebo for six menstrual cycles. At the onset of PMDD symptoms, participants will take two pills of their assigned treatment daily. Once symptoms have dissipated, usually around the first or second day of the menstrual cycle, participants will stop taking their assigned treatment for that cycle. For the next 4 months, participants will attend study visits on the fifth day of each monthly menstrual cycle. For the following 2 months, participants will be contacted by telephone. Participants will be asked to rate their mood and symptoms at each contact. A final study visit will be scheduled on the first day of the seventh menstrual cycle. At this point, all participants will be offered sertraline for an additional three menstrual cycles, dosed on a daily basis. Two study visits will be scheduled over the course of the three cycles to evaluate the effectiveness of sertraline when dosed continuously. Urine collection and pregnancy tests may occur at selected times during the study.

ELIGIBILITY:
Inclusion Criteria:

* Menstruating and has cycles between 21 and 35 days
* Meets DSM-IV criteria for PMDD
* Experienced symptoms of PMDD in at least 9 of 12 menstrual cycles within 1 year of study entry
* Willing to use an effective form of birth control throughout the study

Exclusion Criteria:

* Meets MINI DSM-IV criteria for major depressive episode, substance abuse, bulimia nervosa, anorexia, bipolar disorder, or a psychotic disorder, such as schizophrenia or schizoaffective disorder, within 6 months of study entry
* Meets MINI DSM-IV criteria for a substance dependence disorder within 12 months of study entry
* Shows follicular phase symptoms consistent with a diagnosis of major depression
* Shows symptoms consistent with bipolar disorder
* Diagnosed with a severe, clinically significant co-existing condition that may prevent study participation
* Suicidal
* Taking ongoing antidepressant or other psychotropic medication
* History of hypersensitivity or an adverse reaction to sertraline
* Pregnant or breastfeeding
* Currently undergoing treatment with a depot hormonal preparation or any other medication that would lead to a lack of menses or markedly irregular menses
* Using a hormonal contraceptive pill or hormonal device within 6 months of study entry
* Taking a hormonal contraceptive pill that includes 20 micrograms of ethinyl estradiol and 3 micrograms of drospirenone
* Has been in individual psychotherapy or individual counseling for 3 months or less at study entry

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Actual)
Dates: Start 2007-11-06 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A. Yonkers, MD, Principal Investigator — Yale University; Margaret Altemus, MD, Principal Investigator — Weill Medical College of Cornell University; Susan Kornstein, MD, Principal Investigator — Virginia Commonwealth University School of Medicine
Locations (3):
- United States (3):
  - Yale University School of Medicine, New Haven, Connecticut
  - Cornell University, Weill Medical College, New York, New York
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No
we will share data with a data request that is reviewed by investigators

REFERENCES:
- [Background] Yonkers KA, O'Brien PM, Eriksson E. Premenstrual syndrome. Lancet. 2008 Apr 5;371(9619):1200-10. doi: 10.1016/S0140-6736(08)60527-9. PMID 18395582
- [Background] Wallenstein GV, Blaisdell-Gross B, Gajria K, Guo A, Hagan M, Kornstein SG, Yonkers KA. Development and validation of the Premenstrual Symptoms Impact Survey (PMSIS): a disease-specific quality of life assessment tool. J Womens Health (Larchmt). 2008 Apr;17(3):439-50. doi: 10.1089/jwh.2007.0377. PMID 18328013
- [Background] Borenstein JE, Dean BB, Leifke E, Korner P, Yonkers KA. Differences in symptom scores and health outcomes in premenstrual syndrome. J Womens Health (Larchmt). 2007 Oct;16(8):1139-44. doi: 10.1089/jwh.2006.0230. PMID 17937566
- [Background] Borenstein JE, Dean BB, Yonkers KA, Endicott J. Using the daily record of severity of problems as a screening instrument for premenstrual syndrome. Obstet Gynecol. 2007 May;109(5):1068-75. doi: 10.1097/01.AOG.0000259920.73000.3b. PMID 17470584
- [Background] Halbreich U, Backstrom T, Eriksson E, O'brien S, Calil H, Ceskova E, Dennerstein L, Douki S, Freeman E, Genazzani A, Heuser I, Kadri N, Rapkin A, Steiner M, Wittchen HU, Yonkers K. Clinical diagnostic criteria for premenstrual syndrome and guidelines for their quantification for research studies. Gynecol Endocrinol. 2007 Mar;23(3):123-30. doi: 10.1080/09513590601167969. PMID 17454164
- [Result] Hartlage SA, Freels S, Gotman N, Yonkers K. Criteria for premenstrual dysphoric disorder: secondary analyses of relevant data sets. Arch Gen Psychiatry. 2012 Mar;69(3):300-5. doi: 10.1001/archgenpsychiatry.2011.1368. PMID 22393222
- [Derived] Yonkers KA, Altemus M, Gilstad-Hayden K, Kornstein SG, Gueorguieva R. Does Symptom-Onset Treatment With Sertraline Improve Functional Impairment for Individuals With Premenstrual Dysphoric Disorder?: A Randomized Controlled Trial. J Clin Psychopharmacol. 2023 Jul-Aug 01;43(4):320-325. doi: 10.1097/JCP.0000000000001700. Epub 2023 May 22. PMID 37212651
- [Derived] Yonkers KA, Kornstein SG, Gueorguieva R, Merry B, Van Steenburgh K, Altemus M. Symptom-Onset Dosing of Sertraline for the Treatment of Premenstrual Dysphoric Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Oct;72(10):1037-44. doi: 10.1001/jamapsychiatry.2015.1472. PMID 26351969
- See also: Click here for the PMS, Perinatal, and Postpartum Research Program's Web site — http://www.researchforher.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three-center study; New Haven, CT; New York City, NY; Richmond, VA. Participants recruited via direct mail and advertisements. Assessed initially over phone, then face-to-face screening office visit. Screening took place between September 2007 and February 2012.
Groups:
- Sertraline: Participants will take sertraline that is dosed between 50 and 100 mgs during the symptomatic period
  Sertraline: 50 mg of sertraline will be taken at the onset of premenstrual symptoms through the first few days of menses. If a participant shows an insufficient response to this dose, the dose may be increased to 100 mg. Women who report moderate to severe side effects will be allowed to reduce their dose to 25 mg of sertraline and to increase the dose at the next cycle unless rate-limiting side effects continue.
- Placebo: Participants will take similarly looking placebo during the symptomatic period
  Placebo: 50 mg of placebo will be taken at the onset of premenstrual symptoms through the first few days of menses. If a participant shows an insufficient response to this dose, the dose may be increased to 100 mg.
Period: Overall Study
Arm/Group | Sertraline | Placebo
Started | 125 | 127
Cycle 1 | 110 | 123
Cycle 2 | 104 | 112
Cycle 3 | 100 | 101
Cycle 4 | 95 | 98
Cycle 5 | 88 | 85
Cycle 6 | 88 | 88
Completed | 88 | 88
Not Completed | 37 | 39
Not completed — Lost to Follow-up | 15 | 14
Not completed — Withdrawal by Subject | 16 | 12
Not completed — Adverse Event | 2 | 2
Not completed — Rescue | 3 | 9
Not completed — Pregnancy | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis included all women enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline | Placebo | Total
Number analyzed (Participants) | 125 | 127 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] — mean age in years
  years | 33.7 (6.71) | 34.6 (6.90) | 34.17 (6.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 127 | 252
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 86 | 89 | 175
  Black | 19 | 20 | 39
  Hispanic | 15 | 13 | 28
  Asian/mixed/other | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 125 | 127 | 252
Education [Number; unit: participants]
  Missing | 1 | 0 | 1
  Some high school/high school graduate | 11 | 11 | 22
  Some college | 40 | 22 | 62
  College/graduate or professional school | 73 | 94 | 167
Marital status [Number; unit: participants]
  Married | 51 | 42 | 93
  Living with partner | 14 | 20 | 34
  Divorced/separated | 11 | 14 | 25
  Never married | 49 | 51 | 100
Past Psychiatric Conditions: Major Depressive Disorder [Number; unit: participants]
  Yes | 35 | 43 | 78
  No | 90 | 84 | 174
Baseline Length of Menstrual Cycle [Mean (Standard Deviation); unit: days] | 27.92 (5.26) | 27.02 (4.58) | 27.4 (4.9)
Baseline Luteal Phase Daily Rating of Severity of Problems Score [Mean (Standard Deviation); unit: units on a scale] — Daily Rating of Severity of Problems (DRSP), composed of 21 items reflecting 11 candidate symptoms for PMDD each scored 1-6. Min=11 (asymptomatic), Max=66 (Highly symptomatic), higher scores indicate most severe problems
  units on a scale | 61.20 (20.09) | 60.37 (17.37) | 60.8 (18.7)

OUTCOME MEASURES:

1. Primary Outcome: Premenstrual Tension Scale (PMTS)
Description: The PMTS is a 10-item scale constructed to study premenstrual syndromes. It is sensitive to change with treatment. It includes items of irritability-hostility, tension, efficiency, dysphoria, motor coordination, mental-cognitive functioning, eating habits, social impairment, sex drive, and physical symptoms. PMTS-O or PMTS-SR? Min=0 (asymptomatic), Max=40 (Highly symptomatic), higher scores indicate most severe problems
Time Frame: Measured from baseline to Cycle 6
Population: all randomized participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 125 | 127
units on a scale
  Baseline | 22.3 (4.8) | 21.4 (4.5)
  Cycle 1 | 15.6 (7.3) | 16.8 (6.0)
  Cycle 2 | 14.1 (6.9) | 15.6 (6.1)
  Cycle 3 | 13.0 (8.0) | 14.0 (5.8)
  Cycle 4 | 12.9 (6.7) | 13.9 (6.3)
  Cycle 5 | 11.4 (6.3) | 12.4 (6.3)
  Cycle 6 | 11.7 (6.8) | 12.8 (6.9)
  Average change from baseline | -10.6 (6.6) | -8.9 (7.4)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Group comparison; Test type: Superiority or Other; p = 0.21, ANOVA
Statistical Analysis 2: Comparison: Sertraline vs Placebo; Change over time in both groups; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Sertraline vs Placebo; Group by time: comparison of rates of change; Test type: Superiority or Other; p = 0.06, ANOVA
Statistical Analysis 4: Comparison: Sertraline vs Placebo; Estimated mean difference from baseline to endpoint between active vs. placebo; Test type: Superiority or Other; p = 0.049, Mixed Models Analysis; Mean Difference (Net) = 1.88, 95% CI 2-sided [0.01 to 3.75], Standard Error of Mean 0.95

2. Primary Outcome: Inventory of Depression Symptoms (IDS-C)
Description: Inventory of Depressive Symptomatology-Clinician version (IDS-C) - a depression measure that has 28 items and detects appropriate variations between follicular and luteal phases in subjects with PMDD. Min score is 0, max is 84.Lower score is less symptomatic.
Time Frame: Measured from baseline to Cycle 6
Population: all participants enrolled were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 125 | 127
units on a scale
  Baseline | 35.4 (10.7) | 32.8 (10.4)
  Cycle 1 | 23.7 (12.3) | 24.0 (11.4)
  Cycle 2 | 21.0 (11.7) | 22.8 (10.6)
  Cycle 3 | 19.2 (13.1) | 19.6 (10.0)
  Cycle 4 | 17.3 (11.1) | 19.1 (9.9)
  Cycle 5 | 15.2 (9.9) | 16.7 (10.4)
  Cycle 6 | 15.5 (10.7) | 17.8 (11.0)
  Average change from baseline | -20.0 (11.4) | -15.3 (12.5)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Group comparison; Test type: Superiority or Other; p = 0.54, ANOVA
Statistical Analysis 2: Comparison: Sertraline vs Placebo; Change over time in both groups; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Sertraline vs Placebo; Group by time: comparison of rates of change; Test type: Superiority or Other; p = 0.02, ANOVA
Statistical Analysis 4: Comparison: Sertraline vs Placebo; Estimated mean difference from baseline to end point between active vs. placebo; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis; Mean Difference (Net) = 5.14, 95% CI 2-sided [1.97 to 8.31], Standard Error of Mean 1.62

3. Primary Outcome: Michelson SSRI Withdrawal Checklist
Description: Michelson SSRI Withdrawal Checklist - 16-item (not exactly 17-item, mood swings and crying were in DRSP) including dizziness, nausea, unusual dreams, chills, increased sweating, loose stools, agitation, ringing or noises in the ears. Items were summed for 3 days after pill-taking ended for each menstrual cycle.Scale is 0-80 for total range of the scale with lower less severe. There are no units
Time Frame: Measured from Cycle 1 to Cycle 6
Population: all participants enrolled were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 125 | 127
units on a scale
  Cycle 1 | 72.9 (29.3) | 68.1 (25.4)
  Cycle 2 | 73.4 (29.9) | 75.2 (33.1)
  Cycle 3 | 70.3 (27.9) | 71.7 (39.0)
  Cycle 4 | 62.3 (25.1) | 65.4 (25.3)
  Cycle 5 | 63.9 (19.9) | 62.1 (24.0)
  Cycle 6 | 67.5 (22.1) | 76.2 (34.1)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Group comparison; Test type: Superiority or Other; p = 0.46, ANOVA
Statistical Analysis 2: Comparison: Sertraline vs Placebo; Change over time in both groups; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Sertraline vs Placebo; Group by time: comparison rates of change; Test type: Superiority or Other; p = 0.69, ANOVA
Statistical Analysis 4: Comparison: Sertraline vs Placebo; Estimated mean difference from Cycle 1 to end point between active vs. placebo; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis; Mean Difference (Net) = 1.02, 95% CI 2-sided [0.83 to 1.26]

4. Secondary Outcome: Clinical Global Severity (CGI-S)
Description: Clinical Global Impressions-Severity is measured on a scale of 1-7, with 7 as most severe.
Time Frame: Baseline through Cycle 6
Population: all participants enrolled analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 125 | 127
units on a scale
  Baseline | 4.5 (0.7) | 4.5 (0.6)
  Cycle 1 | 3.4 (1.0) | 3.8 (0.9)
  Cycle 2 | 3.1 (1.2) | 3.3 (1.1)
  Cycle 3 | 2.8 (1.3) | 3.0 (1.0)
  Cycle 4 | 2.6 (1.2) | 2.9 (1.2)
  Cycle 5 | 2.4 (1.0) | 2.7 (1.1)
  Cycle 6 | 2.2 (1.1) | 2.5 (1.3)
  Average change from baseline | -2.3 (1.2) | -1.9 (1.4)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Group comparison; Test type: Superiority or Other; p = 0.01, Chi-squared
Statistical Analysis 2: Comparison: Sertraline vs Placebo; Change over time in both groups; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Sertraline vs Placebo; Group by time: comparison rates of change; Test type: Superiority or Other; p = 0.28, Chi-squared
Statistical Analysis 4: Comparison: Sertraline vs Placebo; Estimated mean difference from baseline to end point between active vs. placebo; Test type: Superiority or Other; p = 0.056, Mixed Models Analysis; Mean Difference (Net) = 0.59, 95% CI 2-sided [0.30 to 1.19]

5. Other Pre Specified Outcome: Adverse Events
Description: A measurement of frequency of adverse events by random assignment
Time Frame: Baseline through Cycle 6
Population: all enrolled participants were analyzed
Measure: Number; unit: participants
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 125 | 127
participants
  Nausea | 15 | 35
  Diarrhea | 14 | 22
  Headache | 19 | 14
  Insomnia | 9 | 22
  Fatigue | 14 | 15
  Mouth dryness | 5 | 13
  Difficulty concentrating | 9 | 8
  Anxiety, agitation | 6 | 10
  Diaphoresis | 10 | 6
  Dizziness/lightheadedness | 6 | 9

6. Primary Outcome: Number of Days Pills Were Taken
Description: The number of days that pills were taken on.
Time Frame: Measured from Cycle 1 to Cycle 6
Population: all participants enrolled were analyzed
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 125 | 127
number of days
  Cycle 1 | 6.5 (3.4) | 6.6 (3.4)
  Cycle 2 | 7.4 (3.3) | 6.7 (3.3)
  Cycle 3 | 8.2 (3.7) | 7.1 (3.4)
  Cycle 4 | 7.0 (3.8) | 6.9 (3.4)
  Cycle 5 | 7.6 (4.0) | 6.7 (3.4)
  Cycle 6 | 6.9 (3.8) | 6.1 (3.7)
  Average Change from Cycle 1 | 0.3 (4.2) | -0.3 (3.6)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Group comparison; Test type: Superiority or Other; p = 0.30, ANOVA
Statistical Analysis 2: Comparison: Sertraline vs Placebo; Change over time in both groups; Test type: Superiority or Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Sertraline vs Placebo; Group by time: comparison rates of change; Test type: Superiority or Other; p = 0.73, ANOVA
Statistical Analysis 4: Comparison: Sertraline vs Placebo; Estimated mean difference from baseline to end point between active vs. placebo; Test type: Superiority or Other; p = 0.06, Mixed Models Analysis; Mean Difference (Net) = 1.12, 95% CI 2-sided [0.92 to 1.35]

7. Primary Outcome: Number of Symptomatic Days Before Pills Were Taken
Description: Symptomatic days were those that participant experienced at least 3 symptoms at a severity of at least "3", which is a mean of at least mild.
Time Frame: Cycle 1 to Cycle 6
Population: all enrolled participants were analyzed
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 125 | 127
days
  Cycle 1 | 2.8 (3.0) | 2.6 (3.0)
  Cycle 2 | 2.0 (2.2) | 2.7 (3.1)
  Cycle 3 | 1.9 (2.8) | 2.0 (2.7)
  Cycle 4 | 2.0 (2.7) | 2.0 (2.9)
  Cycle 5 | 1.9 (2.9) | 1.8 (2.4)
  Cycle 6 | 1.7 (2.3) | 2.0 (3.2)
  Average Change from Cycle 1 | -0.7 (3.4) | -1.0 (3.2)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Group comparison; Test type: Superiority or Other; p = 0.80, ANOVA
Statistical Analysis 2: Comparison: Sertraline vs Placebo; Change over time in both groups; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Sertraline vs Placebo; Group by time: comparison rates of change; Test type: Superiority or Other; p = 0.43, ANOVA
Statistical Analysis 4: Comparison: Sertraline vs Placebo; Estimated mean difference from baseline to endpoint between active vs. placebo; Test type: Superiority or Other; p = 0.61, Mixed Models Analysis; Mean Difference (Net) = 1.11, 95% CI 2-sided [0.85 to 1.45]

8. Primary Outcome: DRSP
Description: DRSP (Daily Rating of Severity Problems) is composed of 21 items reflecting the 11 candidate symptoms for PMDD according to DSM IV and DSM V. Each symptom is scored 1-6. A diagnosis of PMDD requires a minimum average luteal phase score of greater than or equal to 3 (mild) for at least 5 PMDD symptoms during the five most symptomatic of the final seven luteal phase days and the first two days of menses onset, and we require that the average follicular phase score not be >2 on these same items. The minimum score is 0 and maximum is 126 for the total score. A higher score indicates greater severity of symptoms.
Time Frame: Baseline to Cycle 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 113 | 115
units on a scale
  Baseline | 60.3 (19.5) | 59.5 (17.3)
  Cycle 1 | 43.7 (17.4) | 46.1 (17.2)
  Cycle 2 | 38.7 (15.8) | 44.4 (17.5)
  Cycle 3 | 36.8 (15.7) | 40.7 (14.7)
  Cycle 4 | 35.3 (12.2) | 36.9 (11.3)
  Cycle 5 | 31.7 (10.5) | 35.2 (12.7)
  Cycle 6 | 32.2 (10.4) | 36.1 (13.6)
  Average change from baseline | -29.7 (18.8) | -22.4 (16.0)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Group comparison; Test type: Superiority or Other; p = 0.83, ANOVA
Statistical Analysis 2: Comparison: Sertraline vs Placebo; Change over time in both groups; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Sertraline vs Placebo; Group by time: comparison rates of change; Test type: Superiority or Other; p = 0.02, ANOVA
Statistical Analysis 4: Comparison: Sertraline vs Placebo; Estimated mean difference from baseline to end point between active vs. placebo; Test type: Superiority or Other; p = 0.169, Mixed Models Analysis; Mean Difference (Net) = 1.09, 95% CI 2-sided [0.96 to 1.25]

9. Secondary Outcome: DRSP Depression Subscale
Description: Depressive symptoms included: felt depressed, felt hopeless, felt worthless or guilt, slept more, trouble sleeping, felt overwhelmed. Symptoms were scored on a scale of 1-6 The score range is 0-36 with higher indicating greater severity.
Time Frame: Baseline to Cycle 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 113 | 115
units on a scale
  Baseline | 7.5 (4.0) | 7.2 (3.5)
  Cycle 1 | 5.5 (3.0) | 5.7 (8.4)
  Cycle 2 | 4.8 (2.7) | 4.9 (2.4)
  Cycle 3 | 4.6 (2.7) | 4.6 (2.0)
  Cycle 4 | 4.3 (1.9) | 4.3 (1.5)
  Cycle 5 | 3.9 (1.6) | 4.2 (1.8)
  Cycle 6 | 3.9 (2.0) | 4.2 (2.0)
  Average change from baseline | -4.0 (4.0) | -2.7 (3.0)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Group comparison; Test type: Superiority or Other; p = 0.37, ANOVA
Statistical Analysis 2: Comparison: Sertraline vs Placebo; Change over time in both groups; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Sertraline vs Placebo; Group by time: comparison rates of change; Test type: Superiority or Other; p = 0.73, ANOVA
Statistical Analysis 4: Comparison: Sertraline vs Placebo; Estimated mean difference from baseline to end point between active vs. placebo; Test type: Superiority or Other; p = 0.13, Mixed Models Analysis; Mean Difference (Net) = 1.08, 95% CI 2-sided [0.91 to 1.28]

10. Secondary Outcome: DRSP Physical Subscale
Description: Physical symptoms included breast tenderness, bloating, headache, joint or muscle pain. Symptoms were scored on a scale of 1-6. The severity range is 0-24 with 24 being more symptomatic.
Time Frame: Baseline to Cycle 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 113 | 115
units on a scale
  Baseline | 10.6 (3.6) | 10.6 (3.9)
  Cycle 1 | 8.4 (3.5) | 8.4 (3.6)
  Cycle 2 | 8.2 (3.7) | 8.8 (3.8)
  Cycle 3 | 7.8 (3.2) | 8.1 (3.4)
  Cycle 4 | 7.4 (3.2) | 7.3 (2.8)
  Cycle 5 | 6.9 (2.7) | 7.1 (3.0)
  Cycle 6 | 6.9 (2.6) | 7.4 (2.9)
  Average change from baseline | -4.2 (3.8) | -2.9 (3.5)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Group comparison; Test type: Superiority or Other; p = 0.31, ANOVA
Statistical Analysis 2: Comparison: Sertraline vs Placebo; Change over time in both groups; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Sertraline vs Placebo; Group by time: comparison rates of change; Test type: Superiority or Other; p = 0.46, ANOVA
Statistical Analysis 4: Comparison: Sertraline vs Placebo; Estimated mean difference from baseline to end point between active vs. placebo; Test type: Superiority or Other; p = 0.94, Mixed Models Analysis; Mean Difference (Net) = 1.09, 95% CI 2-sided [0.96 to 1.23]

11. Secondary Outcome: DRSP Anger/Irritability Subscale
Description: Anger/irritability included anger/irritability and conflicts with people. Symptoms were scored on a scale 1-6. The range is 0 to 12 with a higher score indicating greater symptom severity.
Time Frame: Baseline to Cycle 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 113 | 115
units on a scale
  Baseline | 6.4 (2.2) | 6.3 (2.1)
  Cycle 1 | 4.1 (1.9) | 4.6 (2.1)
  Cycle 2 | 3.5 (1.7) | 4.5 (2.3)
  Cycle 3 | 3.3 (1.7) | 4.0 (1.9)
  Cycle 4 | 3.2 (1.4) | 3.8 (1.6)
  Cycle 5 | 2.9 (1.3) | 3.5 (1.7)
  Cycle 6 | 2.8 (1.4) | 3.5 (1.5)
  Average change from baseline | -3.7 (2.2) | -2.8 (1.9)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Group comparison; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Sertraline vs Placebo; Change over time in both groups; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Sertraline vs Placebo; Group by time: comparison rates of change; Test type: Superiority or Other; p < 0.01, ANOVA
Statistical Analysis 4: Comparison: Sertraline vs Placebo; Estimated mean difference from baseline to end point between active vs. placebo; Test type: Superiority or Other; p = 0.027, Mixed Models Analysis; Median Difference (Net) = 1.22, 95% CI 2-sided [1.05 to 1.41]

12. Secondary Outcome: Clinical Global Impressions-Improvement (CGI-I)
Description: The Clinical Global Impressions-Improvement (CGI-I) scale is a 7-point scale with 7 being the least improvement.
Time Frame: Cycle 1 to Cycle 6
Population: all participants who were measured at a visit past baseline were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 110 | 123
units on a scale
  Cycle 1 | 2.7 (1.1) | 3.2 (1.0)
  Cycle 2 | 2.4 (1.0) | 2.7 (1.1)
  Cycle 3 | 2.3 (1.3) | 2.4 (1.0)
  Cycle 4 | 2.1 (1.2) | 2.5 (1.3)
  Cycle 5 | 2.0 (1.0) | 2.1 (1.2)
  Cycle 6 | 1.8 (0.9) | 2.2 (1.3)
  Average change from Cycle 1 | -0.9 (1.2) | -0.8 (1.4)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Group comparison; Test type: Superiority or Other; p = 0.01, Chi-squared
Statistical Analysis 2: Comparison: Sertraline vs Placebo; Group by time: comparison rates of change; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Sertraline vs Placebo; Estimated mean difference between active and placebo groups at end-point only; Test type: Superiority or Other; p = 0.056, Mixed Models Analysis; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [0.30 to 1.02]

ADVERSE EVENTS:
Time Frame: The adverse event data was collected for all participants at each visit. The first visits were in November of 2007 and the trial ended in July of 2012. Adverse event data spanned that 4 and a half year time frame.
Arm/Group | Sertraline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/127
Other Adverse Events (participants affected / at risk) | 48/125 | 40/127
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=125) | Placebo (N=127)
Nausea (Gastrointestinal disorders) | 15 (15) | 35 (35)
Diarrhea (Gastrointestinal disorders) | 14 (14) | 22 (22)
Headache (General disorders) | 19 (19) | 14 (14)
Insomnia (General disorders) | 9 (9) | 22 (22)
Fatigue (General disorders) | 14 (14) | 15 (15)
Mouth Dryness (General disorders) | 5 (5) | 13 (13)
Difficulty Concentrating (General disorders) | 9 (9) | 8 (8)
Anxiety, Agitation (Psychiatric disorders) | 6 (6) | 10 (10)
Diaphoresis (General disorders) | 10 (10) | 6 (6)
Dizziness/lightheadedness (General disorders) | 6 (6) | 9 (9)

LIMITATIONS AND CAVEATS:
Limitations of this study include attrition over time and the restricted dose range of 25-100mg sertraline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No